CLINICAL TRIAL: NCT05570435
Title: Evaluate Efficacy of Milk Product Supplemented With Bioactives in Lowering Post Meal Glucose Response: an Acute Study in Chinese Population
Brief Title: Efficacy of Milk Product Supplemented With Bioactives in Lowering Post Meal Glucose Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 21.16.NR
Record Dates: First submitted 2022-09-20; First posted 2022-10-06 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Healthy; PreDiabetes; Adult; Asian
Keywords: Nestle, postprandial glucose, incretins, insulin, healthy
MeSH Terms: conditions — Prediabetic State; Insulin Resistance | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YIYANG TangLv milk powder (Experimental): 30g of milk powder (Nestle YIYANG TangLv milk powder) containing 789 mg Reducose® extract, standardized to contain 1% 1-deoxynojirimycin (1-DNJ), 10% of an oil mix and 8% of soluble fiber reconstituted with 180 ml of warm water.
  Interventions: Biological: Blood collection
- skimmed milk (Active Comparator): 25g of commercially available skimmed milk powder reconstituted with 180 ml of warm water.
  Interventions: Biological: Blood collection

INTERVENTIONS:
Biological: Blood collection — Blood collection for glucose, insulin, GLP-1, GIP and C-peptide.

SUMMARY:
This is a monocentric, randomized controlled, open-label, 2x2 cross-over study. The main objective of the study is to Evaluate the efficacy of Nestle YIYANG TangLv milk powder in lowering the Post Prandial Glucose Response (PPGR) of a high carbohydrate meal when consumed with the meal.

DETAILED DESCRIPTION:
This is an acute, monocentric, open label, randomized, 2-arm, cross-over, clinical trial in 30 subjects of Chinese Han ethnicity. Subjects will receive the two different interventions in a randomized order. This study will assess the efficacy of the investigational product after a single consumption. Day before (V1 and V3) the intervention visits (V2 and V4) the subjects will be admitted at the investigational site for an overnight stay where they will consume a standardized dinner. V2 and V3 will be followed by a wash-out period of 3 days. The two arms are:

Arm 1: skimmed milk (control) Arm 2: Nestle YIYANG TangLv milk powder

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign written informed consent prior to trial entry
2. Deemed able to comply with study protocol for 2-3 weeks
3. Male or female aged 45-75 years (inclusive 45 and 75)
4. HbA1c test results < 6.5% at Visit 1 (Admission 1)
5. Waist circumference ≤90 cm in males and ≤ 85 cm in females
6. Chinese Han ethnic group
7. BMI >18.5 and <28 kg/m2

Exclusion Criteria:

1. Pre-existing chronic medical or psychiatric conditions, as diagnosed by the treating physician (psychiatric illness, asthma or chronic lung disease requiring long term medications or oxygen, diabetes mellitus, chronic infective disease, including tuberculosis, hepatitis B and C, and HIV)
2. Significant medical or surgical event in the past 3 months potentially interfering with study procedures and assessments
3. Known food allergy in particular cow's milk protein allergy (CMPA), lactose and /or soy intolerance or known hypersensitivity/intolerance to any other ingredients in the study product
4. Known substance abuse or alcohol user exceeds following intake, alcohol intake > 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer
5. Consumption of tobacco products, smoking or chewing tobacco
6. History of significant organ dysfunction or disease
7. Subjects with refractory hypertension, and patients with hypertension who are taking antihypertensive drugs (beta-blockers, thiazide diuretics, etc.) that may affect blood glucose metabolism
8. Females currently on hormonal therapy including post-menopausal hormone replacement therapy (PRT) or have been on PRT treatment in the past two months before study participation
9. Known autoimmune and/or genetic disease
10. Known chronic diarrhea or gastrointestinal discomfort
11. Known endocrine and metabolic diseases under drug treatment (e.g., pituitary tumors, thyrotoxicosis due to various causes, Cushing's syndrome etc.)
12. Subjects on systemic corticosteroids, glucocorticoids, or cyclosporine A
13. Recent blood donation (<8 weeks)
14. Pregnant or lactating women

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
3h-iAUC of PPGR | 3 hours
  Incremental area under the curve (3h-iAUC0-3h) of the post-prandial plasma glucose concentration (PPGR)

SECONDARY OUTCOMES:
iAUC of PPGR | 1hour, 2 hours
  Incremental area under the curve of PPGR (Postprandial Glucose Response)
Tmax of PPGR | 3 hours
  Tmax(the time when Cmax is achieved) of PPGR (Postprandial Glucose Response)
Cmax of PPGR | 3 hours
  Cmax(maximal value of measured timepoints) of PPGR (Postprandial Glucose Response)
iCmax of PPGR | 3 hours
  iCmax( maximal incremental value ) of PPGR (Postprandial Glucose Response)
iAUC of PPIR | 1 hour, 2 hours
  Incremental area under the curve of PPIR (Postprandial Insulin Response)
Tmax of PPIR | 3 hours
  Tmax(the time when Cmax is achieved) of PPIR (Postprandial Insulin Response)
Cmax of PPIR | 3 hours
  Cmax(maximal value of measured timepoints) of PPIR (Postprandial Insulin Response)
iCmax of PPIR | 3 hours
  iCmax( maximal incremental value ) of PPIR (Postprandial Insulin Response)

OTHER OUTCOMES:
additional endpoints slopes derived from PPGR | 0, 15, 30 min or 1 hour, 2 hours, 3 hours
  additional endpoints slopes derived from PPGR

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Cherta-Murillo A, Xu H, Moullan N, Tadi M, Huang F, Kodakuthumparambil N, Campos VC, Li J, Fu Q, Li Q, Huang H, Rytz A, Darimont C, Chen W. Milk with Mulberry Leaf Extract, Vegetable Oil, and Inulin Reduce Early Glucose and Insulin Response in Healthy Adults in China: Randomized Controlled Trial. J Nutr. 2025 Jul;155(7):2227-2235. doi: 10.1016/j.tjnut.2025.05.036. Epub 2025 May 24. PMID 40419093